CLINICAL TRIAL: NCT02961621
Title: Multi-tasking to Hyper-tasking: Investigating the Impact of Next Generation 911
Acronym: NG911
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Hendrika Meischke, Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00001920
Record Dates: First submitted 2016-11-07; First posted 2016-11-11 (Estimated); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Stress, Psychological
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stress Reduction Training Group (Experimental): This group will complete a 7-week online mindfulness-based resiliency training: Stress Reduction Training for 9-1-1 Telecommunicators
  Interventions: Behavioral: Stress Reduction Training for 9-1-1 Telecommunicators
- Control Group (No Intervention): This group is a wait-list control and will be offered the training after all data collection has been completed.

INTERVENTIONS:
Behavioral: Stress Reduction Training for 9-1-1 Telecommunicators
  Arms: Stress Reduction Training Group

SUMMARY:
Emergency call centers across the country are preparing for the Next Generation 911 (NG911) initiative, which will allow citizens to place 9-1-1 "calls" using digital technologies such as text messaging, email, Skype or instant messaging, and will expand emergency information sources to also include streaming video, photo uploads, and automatic crash notifications. The impact of these new information and communication technologies on those tasked with using them in time-sensitive emergency situations is unknown. Our study is designed to address the following hypotheses: 1) We hypothesize that NG911 implementation will have a significant effect on telecommunicator stress levels and 2) A resiliency training tailored to the needs of telecommunicators will mitigate the impact on NG911 implementation on stress levels. We will test these hypotheses through the following specific aims:

Aim 1: Measure levels of stress, job satisfaction and job performance among 9-1-1 telecommunicators before and after the NG911 implementation.

Aim 2: Develop and test the efficacy of an evidence-based resiliency training and worker support intervention to improve psychological well-being and job performance of 9-1-1 telecommunicators.

Aim 3: Build an ABM tool of 9-1-1 call centers to improve 9-1-1 telecommunicator workforce training and smooth transitions to future call center innovations.

ELIGIBILITY:
Inclusion Criteria:

* subjects must be 9-1-1 telecommunicators (call receivers and dispatchers) who work at participating call centers and consent to participate.

Exclusion Criteria:

* We will exclude subjects who do not consent to participate
* We will exclude subjects who do not confirm that they are 21 or older.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 323 (Actual)
Dates: Start 2015-05-01; Primary Completion 2017-11-01 (Actual); Study Completion 2017-12-15 (Actual)

PRIMARY OUTCOMES:
Calgary Symptoms of Stress Inventory | Baseline, immediately post intervention and 3 months post intervention
  Change in the Calgary Symptoms of Stress Inventory results

CONTACTS AND LOCATIONS:
Overall Officials: Hendrika Meischke, PhD, MPH, Principal Investigator — University of Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kerr DC, Ornelas IJ, Lilly MM, Calhoun R, Meischke H. Participant Engagement in and Perspectives on a Web-Based Mindfulness Intervention for 9-1-1 Telecommunicators: Multimethod Study. J Med Internet Res. 2019 Jun 19;21(6):e13449. doi: 10.2196/13449. PMID 31219045
- [Derived] Meischke H, Lilly M, Beaton R, Calhoun R, Tu A, Stangenes S, Painter I, Revere D, Baseman J. Protocol: a multi-level intervention program to reduce stress in 9-1-1 telecommunicators. BMC Public Health. 2018 May 2;18(1):570. doi: 10.1186/s12889-018-5471-0. PMID 29716576